CLINICAL TRIAL: NCT06352697
Title: Efficacy and Safety of Probiotic Lysate (Postbiotic and Metabiotic) Supplementation in Adults MASLD Patients
Brief Title: Probiotic Lysate (Postbiotic and Metabiotic) Supplementation for Adults MASLD Patients (DELI_MASLD Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Collaborators: Taras Shevchenko National University of Kyiv (Other); Danylo Halytsky Lviv National Medical University (Other); Kyiv City Clinical Endocrinology Center (Other); Center for Innovative Medical Technologies of the National Academy of Sciences of Ukraine (Other); MirImmunoFarm (Unknown); Stellar Biotics (Unknown)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DELI_MASLD
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Dysfunction Associated Steatotic Liver Disease; Steatotic Liver Disease; Hepatic Steatosis
Keywords: Postbiotics; metabiotics; L. rhamnosus; L. delbrueckii; Metabolic Dysfunction Associated Steatotic Liver Disease; fatty liver index; hepatic steatosis index
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic lysate (postbiotic and metabiotc) group (Active Comparator): oral, 2 capsules per day (BID) for 3 month treatment
  Interventions: Dietary Supplement: Probiotic lysate (postbiotic and metabiotc)
- Placebo group (Placebo Comparator): placebo, oral, 2 capsules per day (BID) for 3 month treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic lysate (postbiotic and metabiotc) — Each capsule contains 100 mg of cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023 in powder
  Arms: Probiotic lysate (postbiotic and metabiotc) group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The current study aim was to conduct placebo-controlled randomize clinical trial to assess the short-term efficacy and safety of postbiotics on hepatic fat content as measured by biochemichal hepatic steatosis indeces, serum lipid profile, transaminases activity and chronic systemic inflammatory markers in MASLD patients.

The study will include 3 periods. Screening period of up to 1 weeks to assess the eligibility to inclusion/exclusion criteria. Treatment period for 3 month where the participants will receive a twice daily oral dose of postbiotics (cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023) at the assigned dose of 100mg or placebo in capsules. During this period monthly phone contacts will be done for assessment of compliance and safety concerns. Follow-up period of up to 3 month.

DETAILED DESCRIPTION:
The scientific literature points to the beneficial properties of probiotics in the process of regulating metabolism, yet at the same time, some scientific papers question the effectiveness and the safety of probiotics. In turn, postbiotics and metabiotics are preparations of inanimate microorganisms and / or their components, which are directly identified with the safety of their use and the health benefits of the host. Due to the chemical structure of postbiotics and metabiotics, it is found that they have many health benefits; in particular, they have a local effect on certain tissues of the intestinal epithelium, and influence on many other organs and tissues. It is postbiotics metabolites and metabiotics structural cell fragments that create the appearance of a therapeutic effect of probiotics, which, in turn, limits the risk of introducing living microorganisms into a weakened immune defence. It should also be pointed out that postbiotics and metabiotics are more stable and have a longer shelf-life.

The practical use of probiotics and the study of the mechanism of their action made lately to find that a certain level of biological activity is preserved by dead probiotic cells and even their lysates, which are the natural mixes of metabiotic and postbiotic substances; a biological activity which is strongly oriented toward gut health and immune system regulation. Because probiotic lysates demonstrated biological activity without any of the potential adverse side effects associated with live bacterial cells, one of the future goal is research of the novel postbiotics and metabiotics substances, their individual structures and biological characteristics for understanding their way of communications with host cells and microbiota representatives.

Considering the high biological activity and safety of postbiotics and metabiotic substances, it can be concluded that such a treatment vector will be promising in the near future. That's why our investigation will concentrate on postbiotic, a supplement containing dry fermented cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023.

Recent scientific animal studies on the stated issues point to the benefits of some postbiotics in treating metabolic disorders. The current study aim was to conduct placebo-controlled randomize clinical trial to assess the short-term efficacy and safety of postbiotics on hepatic fat content as measured by biochemichal hepatic steatosis indeces, serum lipid profile, transaminases activity and chronic systemic inflammatory markers in MASLD patients.

The study will include 3 periods. Screening period of up to 1 weeks to assess the eligibility to inclusion/exclusion criteria. Treatment period for 3 month where the participants will receive a twice daily oral dose of postbiotics (cell lysate and DNA fragments of the probiotic strain L. rhamnosus DV - NRRLB-68023) at the assigned dose of 100mg or placebo in capsules. All capsules will be identical with similar organoleptic characteristics (e.g., taste and appearance). Follow-up period of up to 3 month.

The pre-randomization period will be designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study start, after inform consent signed, patients were instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants were instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent the study were instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits were provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy was compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (ages 18-70)
* presence of MASLD according to "A multisociety Delphi consensus statement", 2023;
* the diagnosis of fatty liver was based on the results of abdominal ultrasonography. Of 4 known criteria (hepato-renal echo contrast, liver brightness, deep attenuation, and vascular blurring), the participants were required to have hepato-renal contrast and liver brightness to be given a diagnosis of SLD
* fatty liver index (FLI) more than 60;
* BMI 25-39.9 kg/m2;
* aspartate transaminase (AST) and alanine transaminase (ALT) ≤3x upper limit of normal;
* written informed consent.

Exclusion Criteria:

* recent hepatitis, or positive screening test for hepatitis B (hepatitis B virus surface antigen) or hepatitis C (hepatitis C antibody);
* alcohol abuse (>20 g/day (2 standard drinks) in women or > 30 g/d (3 drinks) in men over a two-year period);
* drug-induced liver disease, Wilson's disease, hereditary deficiency of antitrypsin-1 and idiopathic hemochromatosis;
* history of decompensated liver disease including ascites, encephalopathy or variceal bleeding;
* regular use of an agents with gut microbiota modulation activity (antibiotic, pro-, pre-, post or synbiotics supplement etc.) within 3 months prior to enrollment;
* allergy on probiotics or their components;
* use of agents such as vitamin E, omega-3 fatty acids or medications with evidence for effects on NAFLD (pioglitazone, GLP-1 analogues, dipeptidyl peptidase IV inhibitors, ursodeoxycholic acid);
* subjects with a history of bariatric surgery or significant weight loss (> 5% body weight) or rapid weight loss (> 1.6kg/week), within 6 months prior to enrollment;
* uncontrolled cardiovascular or respiratory disease, decompensated liver disease including ascites, encephalopathy or variceal bleeding, active malignancy, or chronic infections;
* participant who had severe course of COVID-19 (extracorporeal membrane oxygenation, mechanically ventilated), and/or had a confirmed case of COVID-19 within 4 weeks prior to enrollment;
* participation in other clinical trials;
* presence of pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
changes in fatty liver index (FLI) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  FLI = [e 0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (ggt) + 0.053*waist circumference - 15.745) / (1 + e 0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (ggt) + 0.053*waist circumference - 15.745)] × 100
hepatic steatosis index (HSI) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  HSI = 8 x ALT/AST + BMI(+ 2 if type 2 diabetes yes, + 2 if female)
TyG index | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  TyG = ln [Fasting triglyceride (mg / dl) x Fasting glucose (mg / dl)] / 2

SECONDARY OUTCOMES:
Concentration of AST | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  AST in IU/L
Concentration of ALT | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  ALT in IU/L
Concentration of Gamma-glutamyl Transferase (GGT) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  GGT in IU/L
Concentration of Total Cholesterol (TC) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  TC in mmol/l
Concentration of Tryglicerides (TG) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  TG in mmol/l
Concentration of LDL-Cholesterol (LDL-C) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  LDL-C in mmol/l
Concentration of VLDL-Cholesterol (VLDL-C) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  VLDL-C in mmol/L
Concentration of HDL-Cholesterol (HDL-C) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  HDL-C in mmol/L
Concentration of high sensitivity CRP (hs-CRP) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  hs-CRP in mg/L
Concentration of IL-6 | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  IL-6 in pg/mL
waist circumferences (WC) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  WC in cm
body mass index (BMI) | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  weight in kg and height in meters will be combined to report BMI in kg/m^2
visceral fat content | at 3 month (end of treatment) and 6 month (follow-up period) compared to baseline]
  visceral fat content using electronic scales-analyzers of body composition Tanita Scale BC-601

CONTACTS AND LOCATIONS:
Locations (5):
- Ukraine (5):
  - Bogomolets National Medical University, Kyiv
  - Kyiv City Clinical Endocrinology Center, Kyiv
  - Taras Shevchenko National University of Kyiv, Kyiv
  - Center for Innovative Medical Technologies of the National Academy of Sciences of Ukraine, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv

IPD SHARING:
Plan to Share IPD: No